CLINICAL TRIAL: NCT01671137
Title: A Randomized Controlled Trial of Lactobacillus Rhamnosus Strain GG for The Prevention of Functional Abdominal Pain Children After Acute Gastroenteritis
Brief Title: Probiotic for the Prevention of Functional Disorders in Childhood
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Ruggiero Francavilla, MD, PhD, University of Bari
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PrevenDAR; Prevent-001 (Other Grant/Funding Number: Uniba001)
Record Dates: First submitted 2012-08-16; First posted 2012-08-23 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Gastroenteritis
Keywords: Lactobacillus GG; Functional Abdominal Pain; Children; Acute; Gastroenteritis
MeSH Terms: conditions — Gastroenteritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactobacillus Rhamnosus Strain GG (Active Comparator): LGG (6 × 109 colony forming units)
  Interventions: Other: Lactobacillus Rhamnosus Strain GG
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Lactobacillus Rhamnosus Strain GG

INTERVENTIONS:
Other: Lactobacillus Rhamnosus Strain GG — Lactobacillus Rhamnosus Strain GG
  Other Names: LGG

SUMMARY:
The present study has several aims:

1. Establish whether Lactobacillus Rhamnosus Strain GG is able to prevent the onset of IBS in a high risk group of children enrolled after an acute gastroenteritis (the study has been powered to this aim).
2. Establish whether Lactobacillus Rhamnosus Strain GG is able to stabilize the intestinal microbiota after an acute gastroenteritis.
3. Define the intestinal microbiota of children following an acute gastroenteritis and identify, if possible, a modification of the microbiota that can predict the emergence of Irritable Bowel Syndrome.

DETAILED DESCRIPTION:
Study Design A randomized, double-blind, placebo-controlled, parallel-group trial planned following the recommendations established by the Consensus report on clinical trial in IBS.

Children during/after an acute episode of gastroenteritis will enter a 12 months treatment (m1-m12) period followed by a 6 months follow-up phase (m13-m18).

Children will be assigned consecutive numbers, starting with the lowest number available, and randomly assigned, with the use of a computer generated randomisation list using permuted block design, to receive orally either LGG (6 × 109 colony forming units) or placebo (capsules identical in taste and appearance to the active study product except for the absence of LGG) once a day. Enrolled children will be entered sequentially to receive the assigned treatment. Boxes containing placebo will have the same shape, dimension, indication and appearance as those containing the viable LGG and will be provided by the probiotic producer (Dicofarm SpA, Rome, Italy) which ensure that the study is blinded for investigators and patients. Group assignment will be concealed from participants and investigators.

Power calculation With the assumption that, in a 12 month period, IBS would be expected in 16% of children after an episode of acute gastroenteritis as opposed to 5% in the general paediatric population without gastroenteritis, we calculated that a sample of 210 children per group would be required for the study to have 80% power to show an advantage of LGG over placebo in reducing the rate of IBS, based on a two-sided type 1 error rate of 5%..

Eligibility of Patients Patients recruited from primary care paediatricians or paediatric wards during/after (less seven days) an episode of gastroenteritis (bacteria/viruses/parasites).

Inclusion criteria:

1. Children of 2 - 16 years of age;
2. Either sex.

Exclusion criteria:

1. Chronic disease,
2. Clinical history of abdominal pain history suggestive for functional dyspepsia/aerophagia/abdominal migraine
3. Growth failure,
4. Alarm signs of organic conditions.

Assessments, Compliance and Adherence. During the duration of the trial (m1-m18) patients will record gastrointestinal symptoms on monthly bases and the following data will be collected: a) questionnaire of frequency/severity of pain, b) school absence and c) GI symptom score by the compilation of the gastrointestinal symptom rating score.

To assess the severity of pain a combination of the self-report Visual Analogue Scale (VAS) and the Faces Pain Scale (FPS) will be used. The 0-10 mm VAS scale (0 no pain, 10 worst possible pain) included a horizontal colour gradient (green-red), plus a rating. When asked to evaluate pain, the child would point to a level and trace a line. This particular VAS is a validated standard to evaluate pain in children older than five. Assessment was eased coupling the VAS with the FPS that consists of six faces ranging from a relaxed face to a face showing intense pain.

Gastrointestinal symptom rating score (GSRS) consists of a 15-point questionnaire to assess severity and frequency of symptoms validated by Svedlund et al..

During the six months of follow-up the questionnaire will be compiled every other months and the GSRS at month 18.

The impact on parent's overall assessment of treatment will be obtained by a monthly interview by the question "how do you feel the medication is affecting the health of your child?"; possible answers are significant, mild, or no relief.

To ensure compliance one investigator will contact the families every four weeks to monitor the process of the study. Adherence will be measured by counting the number of capsules returned at the study visit; children who missed for more than 20% of the medications were considered noncompliant.

Outcome Measures Primary outcome will be the incidence in IBS in children receiving LGG as compared to those receiving placebo. We have chosen pain as the primary outcome measure, in line with the proposed points-to-consider for IBS trials.

IBS or chronic abdominal pain will be diagnosed and categorised according to ROME III criteria.

Secondary outcomes are: 1) evaluation of frequency/severity of symptoms according to treatment arm; 2) evaluation of perception of children's health according to parents and 3) modification of intestinal microbiota.

Intestinal microbiota The intestinal microbiota will be assesses according to methods published elsewhere.

To define the modification of the intestinal microbiota following an acute gastroenteritis and to determine whether the onset of the IBS is anticipated by a modification of intestinal microbiota we will proceed to the collection of faecal samples at entry, after one month and every two months after enrolment. During the six months of follow-up a fecal sample will be collected only at month 18.

Bacteria DNA in stools will be extracted and stored at -80°C for future analysis. At the end of the trial a subset of informative fecal bacterial DNA will be assessed: a) patients that have NOT developed IBS (LGG and placebo), b) patients that have developed IBS (LGG and placebo).

The analysis of the intestinal microbiota of these informative cases will help to assess whether there is a intestinal microbiota suggestive of future inset of IBS and ability of LGG to stabilize the intestinal microbiota.

Adverse Events and Disallowed Medication Adverse events were monitored throughout the study. Children will not allowed to consume any probiotic other than those provided (except for a transient period no longer that 2 weeks) and they will be invited to continue their eating and physical exercise habits. Concomitant use of medications affecting gastrointestinal motility and/or pain perception was allowed, providing parents registered the intake.

ELIGIBILITY:
Inclusion Criteria:

1. Children of 3 - 16 years of age;
2. Either sex.

Exclusion Criteria:

1. Chronic disease,
2. Clinical history of abdominal pain history suggestive for functional dyspepsia/aerophagia/abdominal migraine
3. Growth failure,
4. Alarm signs of organic conditions.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-07 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Prevention of Abdominal pain | 18 months
  Primary outcome will be the incidence in IBS in children receiving LGG as compared to those receiving placebo. We have chosen pain as the primary outcome measure, in line with the proposed points-toconsider for IBS trials (Corazziari E. Consensus report: Clinical trial guidelines for pharmacological treatment of irritable bowel syndrome. Aliment Pharmcol Ther 2003;18:569).
  IBS or chronic abdominal pain will be diagnosed and categorised according to ROME III criteria (Rasquin A, Di Lorenzo C, Forbes D, et al. Childhood functional gastrointestinal disorders: child/adolescent. Gastroenterology. 2006;130).

SECONDARY OUTCOMES:
Incidence of IBS | 6 months
  Evaluation of frequency/severity of symptoms according to treatment arm;
Children's health | 24 months
  Evaluation of perception of children's health according to parents
Intestinal microbiota | 24 months
  Investigate the modification of intestinal microbiota.

CONTACTS AND LOCATIONS:
Overall Officials: Ruggiero Francavilla, Principal Investigator — University of Bari; Ruggiero FRANCAVILLA, Principal Investigator — DEPARTMENT OF BIOMEDICINA ETA' EVOLUTIVA
Locations (1):
- Clinica Pediatrica, Bari, Apulia, Italy